CLINICAL TRIAL: NCT01032928
Title: Respiratory-Swallow Training in Veterans With Oropharyngeal Cancer
Acronym: RSPT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C7135-R; RX000152-01A1 (Registry Identifier: Dept of Veterans Affairs, ORD)
Record Dates: First submitted 2009-12-14; First posted 2009-12-16 (Estimated); Results first posted 2014-12-04 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2014-12

CONDITIONS: Oropharyngeal Dysphagia; Oropharyngeal Cancer
Keywords: Swallowing; Dysphagia; Breathing and swallowing; Oropharyngeal cancer
MeSH Terms: conditions — Deglutition Disorders; Oropharyngeal Neoplasms; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Respiratory Phase Training (Experimental): Chronically dysphagic, medically stable patients at least 6 months post treatment for head and neck cancer with non-optimal respiratory-swallowing patterns participated in up to 8 sessions of respiratory phase training to learn an optimal respiratory - swallow phase pattern
  Interventions: Behavioral: Respiratory-Swallow Phase training

INTERVENTIONS:
Behavioral: Respiratory-Swallow Phase training — Patients were presented with visually guided respiratory feedback to train optimal respiratory-swallow coordination patterns.

SUMMARY:
Cancers of the head and neck require surgical, radiation, and chemotherapy treatments that are intended to cure the disease. These treatments have toxic effects on muscles and structures that are necessary to swallow safely and efficiently. The resulting swallowing problems (dysphagia) often remain chronic for Veterans and interfere with their ability to eat and drink. The cost burden to the VA health system is high. There is an urgent need to develop rehabilitative treatments that lessen these burdens. The proposed research is designed to test a novel swallowing therapy that includes the coordination of breathing with swallowing. Our study will train medically and surgically treated, chronically dysphagic Veterans with histories of oropharyngeal cancer in a novel therapy that involves both swallowing and respiratory systems. If the therapy is found to be effective, the long term goal of the project is to extend the study to a multi-site, clinical trial and test the longstanding effect of this treatment compared to other swallowing therapies on swallowing function, QOL and cost.

DETAILED DESCRIPTION:
Swallowing impairments (dysphagia) represent the highest functional morbidity in veteran patients treated for oropharyngeal cancers with either surgical approaches followed by radiation or with more recent organ-preservation protocols. The nature of the impairments is often resistive to treatment and results in life-long health consequences and high cost burden on the VA health system. Recent preliminary data have linked alterations in the otherwise highly stable respiratory-swallowing phase pattern relationships to the swallowing impairment and penetration/aspiration and in this patient group. The immediate goal of this clinical trial is to test the effect of a novel respiratory-swallow intervention on swallowing impairment and penetration/aspiration in a cohort of chronically dysphagic veterans following treatment for oropharyngeal cancer. Patients presenting with a "non-optimal" respiratory-swallow phase pattern during liquid swallows and measurable swallowing impairment will learn an "optimal" physiologic pattern that facilitates both airway protective and mechanical advantages during swallowing. The broad goal of this research is to develop ideal respiratory-swallowing phase training methods and regimens that alone or combined with traditional swallowing treatments improve swallowing function in the acute phases of recovery and improve long term patient outcome. Our intention is to use these preliminary data to motivate a larger clinical trial to compare the effect of respiratory-swallow phase training with other evidenced based methods of swallowing treatment and expand the approach to other patient groups that have indications of respiratory-swallow phase impairments (e.g. pulmonary disease and stroke) contributing to impaired swallowing function

ELIGIBILITY:
Inclusion Criteria:

* at least 21 years of age
* agreed to participate in this study and signed an informed consent, either completed by the participant or designated other
* have chronic impairments in oropharyngeal swallowing function following chemotherapy, radiation, and/or surgical intervention for the treatment of first time diagnosis of squamous cell carcinoma of the head and neck
* have completed medical treatments for his/her cancer and any traditional swallowing therapy at least 6 months earlier
* pass a cognitive screening (COGNISTAT)
* have at least one area of impairment (initiation of pharyngeal swallow, anterior hyolaryngeal excursion, extent and duration of PES opening, tongue base retraction, pharyngeal residue) as indicated by the results of the pre-intervention MBSImP (total sum MBSImP
* have PAS scores >/= 3 on 10% of swallows on pre-intervention MBSS
* have a non-optimal (E-I, I-E, or I-I) breathing pattern on 60% of trial swallows.

Exclusion Criteria:

* known allergy or dietary restriction for food or contrast materials used during the exam
* evidence of persistent or recurrent disease on physical examination of the head and neck
* evidence of esophageal stricture noted on MBS
* recurrent oropharyngeal cancer and/or are being treated for other cancer(s) concurrently
* severe COPD (see Pulmonary Criteria below)
* nasogastric feeding tube
* recent change in swallowing status characterized by increase in perceived or observed -swallowing problems by patient, family or testing SLP
* any co-occurring neurological impairment affecting muscle strength and/or cognition
* history of aspiration pneumonia over the past 12 months.
* fail cognitive screening
* absence of swallowing impairment
* evidence of esophageal stricture on MBS
* inability to tolerate at least one of the liquid barium consistencies
* consistent optimal respiratory-swallow phase patterning

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-06; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie J Martin-Harris, Principal Investigator — Ralph H Johnson VA Medical Center, Charleston
Locations (1):
- Ralph H Johnson VA Medical Center, Charleston, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Martin-Harris B, McFarland D, Hill EG, Strange CB, Focht KL, Wan Z, Blair J, McGrattan K. Respiratory-swallow training in patients with head and neck cancer. Arch Phys Med Rehabil. 2015 May;96(5):885-93. doi: 10.1016/j.apmr.2014.11.022. Epub 2014 Dec 11. PMID 25498307
- See also: Click here for more information about this study: Respiratory-Swallow Training in Veterans with Oropharyngeal Cancer — http://www.muschealth.com/ent
- See also: National website for dysphagia research — http://www.dysphagiaresearch.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Head and Neck Clinics at the Ralph H Johnson Veterans Administration Medical Center and the Medical University of South Carolina between May 2010 and April 2013
Pre-assignment Details: 87 participants were recruited; 67 completed screening; 32 were eligible for enrollment; 2 declined participation
Groups:
- Respiratory - Swallow Phase Training: Chronically dysphagic, medically stable patients at least 6 months post treatment for head and neck cancer with non-optimal respiratory-swallowing patterns
Period: Overall Study
Arm/Group | Respiratory - Swallow Phase Training
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Entire Enrolled Study Population
Groups:
- Respiratory-Swallow Phase Training: Chronically dysphagic, medically stable patients at least 6 months post treatment for head and neck cancer with non-optimal respiratory-swallowing patterns
  Respiratory-Swallow Phase training: Will present patients with visually guided, respiratory feedback and train optimal respiratory-swallow coordination patterns, thereby providing the airway protection and mechanical benefits that have been observed in healthy individuals.
Arm/Group | Respiratory-Swallow Phase Training
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Impairment According to the Modified Barium Swallow Impairment Profile (MBSImP)
Description: Analysis of the percentage of impaired swallow components using a dichotomized MBSImP scoring system
Time Frame: Patient were assessed pre-treatment, one week post treatment and one month post treatment. Treatment sessions were twice weekly for up to 4 weeks
Measure: Number; unit: percentage of impairment
Groups:
- Pre-intervention: Subjects eligible for enrollment
- One Week Post Intervention: Subjects that completed treatment were assessed within one week of meeting respiratory-swallow phase training goals
- One Month Post Intervention: VAMC participants were assessed at one month following completion of the treatment protocol
Arm/Group | Pre-intervention | One Week Post Intervention | One Month Post Intervention
Number analyzed (Participants) | 30 | 30 | 15
percentage of impairment
  Lip closure | 5.7 | 9.3 | 2.8
  Tongue control | 58.7 | 53.8 | 59.2
  Bolus transport | 37.3 | 50.2 | 41.5
  Oral residue | 77.3 | 76.4 | 71.1
  Initiation of pharyngeal swallow | 90.4 | 90.8 | 91.1
  Soft palate elevation | 19.8 | 31.0 | 15.6
  laryngeal elevation | 76.6 | 70.8 | 63.3
  Anterior hyiod excursion | 94.7 | 90.5 | 93.3
  Epiglottic inversion | 71.9 | 68.3 | 55.6
  Laryngeal vestibular closure | 78.2 | 55.5 | 62.2
  Pharyngeal stripping wave | 59.3 | 67.6 | 60.7
  Pharyngoesophageal segment opening | 80.6 | 80.5 | 70.0
  Tongue base retraction | 96.0 | 88.6 | 80.7
  Pharyngeal residue | 96.1 | 88.4 | 83.0

2. Secondary Outcome: Percentage of Impairment According to the Penetration-Aspiration Scale
Description: The penetration aspiration scale is a validated 8 point interval scale used to describe penetration and aspiration events. Scores are determined primarily by the depth to which material passes in the airway and by whether or not material entering the airway is expelled. Scores < 3 are considered to be normal. For the purpose of our study scores were dichotimized to normal and impaired.
Time Frame: as for outcome 1
Measure: Number; unit: percentage of swallows with impaired PAS
Arm/Group | Pre-intervention | One Week Post Intervention | One Month Post Intervention
Number analyzed (Participants) | 30 | 30 | 15
percentage of swallows with impaired PAS | 78.0 | 38.3 | 42.2

3. Primary Outcome: Optimal Respiratory - Swallow Phase
Description: Respiratory swallow patterns were collected using nasal airflow and respiratory inductance plethysmography (RIP) of each swallow during the modified barium swallow study. The movements of the ribcage and abdomen were recorded using RIP; data synchronized and recorded using the KayPentax Digital Swallow Workstation Signals Lab. Subjects were categorized as optimal (expiratory-expiratory) versus non-optimal (non-expiratory-expiratory).
Time Frame: as for outcome 1
Measure: Number; unit: percentage of swallows
Groups:
- One Week Post-intervention: Subjects that completed treatment were assessed within one week of meeting respiratory-swallow phase training goals
- One Month Post Intervention: VAMC participants were reassessed at one month post treatment
Arm/Group | Pre-intervention | One Week Post-intervention | One Month Post Intervention
Number analyzed (Participants) | 30 | 30 | 15
percentage of swallows | 43 | 86 | 88.1

ADVERSE EVENTS:
Time Frame: Duration of the study
Description: Patient completed daily EXACT-PRO questionnaires regarding respiratory symptoms. Reported changes were reviewed by pulmonologist
Groups:
- Arm 1: Chronically dysphagic, medically stable patients at least 6 months post treatment for head and neck cancer with non-optimal respiratory-swallowing patterns
  Respiratory-Swallow Phase training: Will present patients with visually guided, respiratory feedback and train optimal respiratory-swallow coordination patterns, thereby providing the airway protection and mechanical benefits that have been observed in healthy individuals.
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes